CLINICAL TRIAL: NCT03420469
Title: Bupropion Stereoselective Disposition and CYP2D6-mediated Drug Interactions in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zeruesenay Desta, Professor of Medicine, Pharmacology and Toxicology, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01GM121707-01A1 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Adverse Effect of Drug Therapy Metabolism Medications (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Bupropion

STUDY DESIGN:
Intervention Model Description: This is an open-label, four-phases, fixed sequence healthy volunteers study investigating: the steady state stereoselective disposition of bupropion and metabolites; and effect of multiple doses of bupropion on CYP2D6 activity, as measured by the metabolism and pharmacokinetics of a single dose of dextromethorphan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baseline CYP2D6 activity (Experimental): CYP2D6 activity will be determined using a single oral dose of dextromethorphan (30 mg PO) as a probe drug at baseline (control).
  Interventions: Drug: Bupropion
- CYP2D6 activity with single dose of bupropion (Experimental): The effect of a single dose of bupropion (150 mg PO) on CYP2D6 activity will be determined using a single oral dose of dextromethorphan (30 mg PO) as a probe drug.
  Interventions: Drug: Bupropion
- CYP2D6 activity after treatment with bupropion to steady sate (Experimental): CYP2D6 activity will be determined using a single oral dose of dextromethorphan (30 mg PO) as a probe drug after 14 days pretreatment with bupropion (150 mg twice daily PO).
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — Phase 1: Baseline CYP2D6 activity, using dextromethorphan (30 mg single dose PO) as a probe drug Phase 2: Single dose bupropion pharmacokinetics and its effect on CYP2D6 activity (determined by dextromethorphan 30 mg single dose PO) Phase 3: Steady state disposition of bupropion and its interaction with CYP2D6 activity (30 mg single dose PO)

SUMMARY:
Primary objectives:

1. To comprehensively characterize steady state stereoselective pharmacokinetics of bupropion and its primary and secondary metabolites in healthy volunteers
2. To prospectively determine the time course (onset), extent and offset of CYP2D6 inhibition in relation to the pharmacokinetic profiles of bupropion and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (approximately 1:1) volunteers between the age of 18 and 55 years old and within 32% of your ideal body weight.
* Judged healthy without any significant medical condition as determined by and decided from a pre-enrollment screening session that include medical history, laboratory tests such as blood and urine tests, and an electrical tracing of the heart beat (electrocardiogram, EKG).
* Individuals who agree to refrain from taking any prescriptions medications, over-the-counter medications, and herbal, dietary, and alternative supplements that may interact with the metabolism of those study drugs at least 2 weeks prior to the start of the study and until study completion.
* Nonsmoker or individuals willing to refrain from smoking or use of tobacco or marijuana for at least two weeks prior to and until the completion of the study (the entire study lasts for approximately 32 days).
* Willing to commit the time requested for this study

Exclusion Criteria:

Subjects will be excluded from the study if they:

* Are underweight (weigh less than 52 kg or 114 lb) or overweight [body mass index (BMI) greater than 32].
* Have laboratory results that do not fall in a healthy range (e.g., blood hemoglobin less than 12.0 mg/dl).
* Have baseline EKG readings that are abnormal that could place the patient at the higher risk as decided by the study medical doctor (MD)
* Have history of intolerance, allergic reactions (e.g. rash) or other forms of hypersensitivities to any of the study medications (dextromethorphan and bupropion).
* Have current alcohol (more than 4 alcoholic drinks per day on a regular basis) or drug abuse.
* Have history or current gastrointestinal (digestive) disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs
* Have history or current seizures, hypertension and heart disease or any other cardiovascular disorders
* Have history or current psychiatric (mental or brain) disorders (e.g., feeling sad or unhappy, loss of interest in normal activities, worried) such as depression, anxiety, or suicidality or suicide attempts.
* Have significantly compromised liver and/or kidney functions.
* Have participated in a research study involving intensive blood sampling or have donated blood within the past two months
* Are unable or unwilling to stop taking other substances that may interfere with the metabolism of the study drugs (bupropion and dextromethorphan) two weeks prior to and during the entire study period, including prescription medications, over-the-counter medications, herbal or dietary supplements, and alternative medicines.
* Are employees or students under supervision of any of the study investigators.
* Cannot state a good understanding of this study including risks and requirements; are unable to follow the rules of this study.
* Cannot commit the time requested for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Exposure | Through study completion, an average of 2 year
  Area under the plasma concentration versus time curves (AUC0-inf) of bupropion and its metabolites as well as CYP2D6 activity measured by dextromethorphan to dextrorphan

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Clinical Research Center (ICRC), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No